CLINICAL TRIAL: NCT03671837
Title: Apneic Oxygenation With a Nasal Cannula in the Obese and Morbidly Obese Surgical Patient: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Apneic Oxygenation With a Nasal Cannula in the Obese and Morbidly Obese Surgical Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tiffany B Moon, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 022017-074
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Apneic; Oxygenation
MeSH Terms: conditions — Apnea | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oyxgen (Experimental): Nasal Insufflation with 15 L/min O2 and a nasopharyngeal airway
  Interventions: Other: Oxygen
- Air (Active Comparator): Nasal Insufflation with 15 L/min air and a nasopharyngeal airway
  Interventions: Other: Air

INTERVENTIONS:
Other: Oxygen — 15 L/min O2
  Arms: Oyxgen
Other: Air — 15 L/min air
  Arms: Air

SUMMARY:
This prospective, randomized, double-blind study is intended to enroll a total of 100 patients with a BMI ≥ 40 kg/m2 and another 100 patients with a BMI ≥ 30 kg/m2 (but less than 40 kg/m2) undergoing surgery with general endotracheal anesthesia at Parkland Hospital. Patients will be randomized to receive either 15 L/min O2 or 15 L/min air from a standard nasal cannula during a simulated prolonged laryngoscopy. The anesthesia provider will do a direct laryngoscopy to ensure that the patient has a Cormack-Lehane grade I-II airway. Patients who have grade III-IV airways will be excluded from further study procedures and not analyzed. The rest of the anesthetic will not deviate from the standard of care. Anesthesia providers will be blinded as to whether patients are receiving oxygen or air during the apneic period.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Obesity (BMI ≥ 30 kg/m2 ≤ 40 kg/m2)
* Morbid obesity (BMI ≥ 40 kg/m2)
* Scheduled for a non-emergent operation that requires general endotracheal anesthesia
* Willing and able to consent in English or Spanish
* No current history of advanced pulmonary or cardiovascular disease

Exclusion Criteria:

* Age less than 18 or older than 70
* BMI < 30 kg/m2
* Patient does not speak English or Spanish
* Family or personal history of malignant hyperthermia
* Patient refusal
* Monitored anesthesia care (MAC) or regional anesthesia planned
* Pregnant or nursing women
* "Stat" (emergent) cases
* Moderate to severe pulmonary disease (e.g., asthma, COPD, pulmonary fibrosis, pulmonary hypertension)
* Respiratory infection within the past 14 days (e.g., pneumonia, bronchitis)
* SpO2 < 97% on room air
* Moderate to severe cardiac disease (e.g., CHF, CAD, aortic stenosis)
* Severe gastroesophageal reflux disease (GERD)
* Nasal obstruction (e.g., tumor)
* Elevated intracranial pressure (e.g., brain tumor)
* History of difficult airway

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Apneic Time | Intraoperative
  To determine whether apneic oxygenation via nasal cannula oxygen results in a longer period of apnea (SpO2 ≥ 95%) during a simulated prolonged laryngoscopy in obese and morbidly obese patients.

SECONDARY OUTCOMES:
Resaturation Time | Intraoperative
  To determine the influence of apneic oxygenation via nasal cannula on the time for resaturation in obese and morbidly obese patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jense HG, Dubin SA, Silverstein PI, O'Leary-Escolas U. Effect of obesity on safe duration of apnea in anesthetized humans. Anesth Analg. 1991 Jan;72(1):89-93. doi: 10.1213/00000539-199101000-00016. PMID 1984382
- [Background] Huang KC, Kormas N, Steinbeck K, Loughnan G, Caterson ID. Resting metabolic rate in severely obese diabetic and nondiabetic subjects. Obes Res. 2004 May;12(5):840-5. doi: 10.1038/oby.2004.101. PMID 15166305
- [Background] McCahon RA, Hardman JG. Fighting for breath: apnoea vs the anaesthetist. Anaesthesia. 2007 Feb;62(2):105-8. doi: 10.1111/j.1365-2044.2007.04932.x. No abstract available. PMID 17223799
- [Background] Baraka AS, Taha SK, Siddik-Sayyid SM, Kanazi GE, El-Khatib MF, Dagher CM, Chehade JM, Abdallah FW, Hajj RE. Supplementation of pre-oxygenation in morbidly obese patients using nasopharyngeal oxygen insufflation. Anaesthesia. 2007 Aug;62(8):769-73. doi: 10.1111/j.1365-2044.2007.05104.x. PMID 17635423
- [Background] Baraka AS, Taha SK, Aouad MT, El-Khatib MF, Kawkabani NI. Preoxygenation: comparison of maximal breathing and tidal volume breathing techniques. Anesthesiology. 1999 Sep;91(3):612-6. doi: 10.1097/00000542-199909000-00009. PMID 10485768
- [Background] Ramachandran SK, Cosnowski A, Shanks A, Turner CR. Apneic oxygenation during prolonged laryngoscopy in obese patients: a randomized, controlled trial of nasal oxygen administration. J Clin Anesth. 2010 May;22(3):164-8. doi: 10.1016/j.jclinane.2009.05.006. PMID 20400000
- [Background] Lopez PP, Stefan B, Schulman CI, Byers PM. Prevalence of sleep apnea in morbidly obese patients who presented for weight loss surgery evaluation: more evidence for routine screening for obstructive sleep apnea before weight loss surgery. Am Surg. 2008 Sep;74(9):834-8. PMID 18807673
- [Background] Heier T, Feiner JR, Lin J, Brown R, Caldwell JE. Hemoglobin desaturation after succinylcholine-induced apnea: a study of the recovery of spontaneous ventilation in healthy volunteers. Anesthesiology. 2001 May;94(5):754-9. doi: 10.1097/00000542-200105000-00011. PMID 11388524
- [Background] Campbell IT, Beatty PC. Monitoring preoxygenation. Br J Anaesth. 1994 Jan;72(1):3-4. doi: 10.1093/bja/72.1.3. No abstract available. PMID 8110546
- [Background] FRUMIN MJ, EPSTEIN RM, COHEN G. Apneic oxygenation in man. Anesthesiology. 1959 Nov-Dec;20:789-98. doi: 10.1097/00000542-195911000-00007. No abstract available. PMID 13825447
- [Background] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Background] Damia G, Mascheroni D, Croci M, Tarenzi L. Perioperative changes in functional residual capacity in morbidly obese patients. Br J Anaesth. 1988 Apr;60(5):574-8. doi: 10.1093/bja/60.5.574. PMID 3377932
- [Background] Don HF, Wahba M, Cuadrado L, Kelkar K. The effects of anesthesia and 100 per cent oxygen on the functional residual capacity of the lungs. Anesthesiology. 1970 Jun;32(6):521-9. doi: 10.1097/00000542-197006000-00012. No abstract available. PMID 5426264
- [Background] Taha SK, Siddik-Sayyid SM, El-Khatib MF, Dagher CM, Hakki MA, Baraka AS. Nasopharyngeal oxygen insufflation following pre-oxygenation using the four deep breath technique. Anaesthesia. 2006 May;61(5):427-30. doi: 10.1111/j.1365-2044.2006.04610.x. PMID 16674614
- [Background] Dyett JF, Moser MS, Tobin AE. Prospective observational study of emergency airway management in the critical care environment of a tertiary hospital in Melbourne. Anaesth Intensive Care. 2015 Sep;43(5):577-86. doi: 10.1177/0310057X1504300505. PMID 26310407
- [Background] Sakles JC, Mosier JM, Patanwala AE, Dicken JM. Apneic oxygenation is associated with a reduction in the incidence of hypoxemia during the RSI of patients with intracranial hemorrhage in the emergency department. Intern Emerg Med. 2016 Oct;11(7):983-92. doi: 10.1007/s11739-016-1396-8. Epub 2016 Feb 4. PMID 26846234